CLINICAL TRIAL: NCT05232318
Title: Apical Root Resorption Accompanied Orthodontic Treatment Using Clear Aligners Versus Fixed Appliances: A CBCT Comparative Study
Brief Title: Root Resorption Accompanied Clear Aligners and Fixed Orthodontic Appliance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Obaida Khaleel Ibrahim, Principal Investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 357/1150
Record Dates: First submitted 2021-12-18; First posted 2022-02-09 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Root Resorption
MeSH Terms: conditions — Root Resorption

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- leveling and alignment using fixed orthodontic appliance (Active Comparator): leveling and alignment using fixed orthodontic appliance
  Interventions: Other: Leveling and alignment
- leveling and alignment using clear aligner (Experimental): leveling and alignment using clear aligner
  Interventions: Other: Leveling and alignment
- leveling and alignment using clear aligner with low level laser therapy (Experimental): leveling and alignment using clear aligner with low level laser therapy
  Interventions: Other: Leveling and alignment

INTERVENTIONS:
Other: Leveling and alignment — Root resorption comparison through the use of CBCT

SUMMARY:
The aim of the study is to compare apical root resorption accompanied orthodontic treatment using clear aligners vs fixed appliances.

DETAILED DESCRIPTION:
by using pretreatment and posttreatment CBCT, root resorption will be measured using a 3D imaging software.

ELIGIBILITY:
Inclusion Criteria:

* Healthy systemic condition/no systemic illness, as reported by patients.
* No use any form of anti - inflammatory drugs the at beginning of study.
* Good oral hygiene.
* Cooperative and motivated.
* In the permanent dentition with all teeth present ( except third molars).
* Minimum to moderate anterior crowding.
* No previous orthodontic treatment.

Exclusion Criteria:

* Previous upper removable orthodontic treatment.
* Patients who required surgery to correct skeletal discrepancies.
* Patients with hyperdontia, hypodontia, or syndromic diseases (e.g. cleft lip and palate).
* Uncooperative patients.
* Patients with poor oral hygiene.

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Amount of Root resorption | 8 months
  Using pretreatment and posttreatment CBCT, volumetric root resorption will be measured by using 3D imaging software

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Abouelnour, Lecturer, Study Director — Lecturer, Department of Orthodontics; Ramadan Y Aboushahba, Associate professor, Study Chair — Associate professor, Department of Orthodontics
Locations (2):
- Egypt (2):
  - AlAzhar Azhar University, Cairo, Or
  - Al Azhar university, Cairo

IPD SHARING:
Plan to Share IPD: No